CLINICAL TRIAL: NCT01659710
Title: Effects of Medical Complexity on the Development of Fidgety Movements and Feasibility of Screening Utilizing the General Movement Assessment for Lurie Children's ICU Patients and Graduates
Brief Title: Effects of Medical Complexity Using GMA on Lurie Children's In- and Outpatients
Acronym: CIMA
Status: Completed | Type: Observational
Sponsor: Raye Ann deRegnier (Other)
Responsible Party: Sponsor-Investigator, Raye Ann deRegnier, Associate Prof of Pediatrics, Ann & Robert H Lurie Children's Hospital of Chicago
Organization: Ann & Robert H Lurie Children's Hospital of Chicago (Other)
Other Study IDs: 2012-14808
Record Dates: First submitted 2012-08-05; First posted 2012-08-08 (Estimated); Last update posted 2024-11-12 (Actual); Status verified 2019-02

CONDITIONS: Medically Complex Infants

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Study Babies: Study video at 50-55 weeks gestational age, motor assessments at 24m (+/- 6 months) and again at 4 years (+/- 1 year).
- Control Babies: Video at 50-55 weeks gestational age, motor assessment at 24 months (+/- 6 months).

SUMMARY:
The purpose of this study is to research a new type of test for cerebral palsy that can be performed earlier, at 10-15 weeks of age (after the due date for premature infants). The test involves a standardized video recording of a baby's natural movements for about 10 minutes. The video recorded movements are evaluated by a special trained observer and also by a computer program. There are some small studies from Europe that suggest that this type of evaluation may be accurate in early diagnosis of cerebral palsy. However, the investigators do not know if this type of evaluation is reliable in large groups of infants, including infants from Children's Memorial Hospital, who tend to be sicker and have more complicated illnesses than many of the European infants. The investigators would therefore like to evaluate whether this type of video recording could be used in the future for early diagnosis of cerebral palsy.

ELIGIBILITY:
Inclusion Criteria:

* Admitted to the NICU/CICU and remain hospitalized at 10-15 weeks postmenstrual age
* Birth at <28 weeks gestation
* Birth weight <1000 grams
* Neurologic risk factors (HIE, abnormal imaging, neonatal seizures, microcephaly)
* Cardiac surgery during first 3 months of life
* Severe chronic lung discharge defined as the need for mechanical ventilation at 36 weeks post-menstrual age
* Discharged home on supplemental oxygen (or if still hospitalized, requiring oxygen at 44 weeks post-menstrual age)

Exclusion Criteria:

* Significant malformations/amputations of the extremities
* Recovering from a surgical procedure within 4 weeks of the assessment
* Physiologic instability precluding movement of the hospital bed or peripheral IV lines that might affect movement of an extremity medication for the purpose of ongoing sedation

Max Age: 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Children's Memorial ICU Patients and Graduates
Sampling Method: Non-Probability Sample
Enrollment: 208 (Actual)
Dates: Start 2012-01 (Actual); Primary Completion 2019-01-31 (Actual); Study Completion 2019-01-31 (Actual)

PRIMARY OUTCOMES:
Presence of cerebral palsy | 24 months (+/- 6 months) and 4 years (+/- 1 year) of age

CONTACTS AND LOCATIONS:
Overall Officials: RayeAnn deRegnier, MD, Principal Investigator — Ann & Robert H Lurie Children's Hospital of Chicago
Locations (1):
- Ann & Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois, United States